CLINICAL TRIAL: NCT01389011
Title: An Evaluation of PI and PVI (Masimo) in Patients With Interscalene Blocks in Orthopedic Surgery
Brief Title: Perfusion Index (PI) and Pleth Variability Index (PVI) in Patients With Interscalene Blocks in Orthopedic Surgery
Acronym: PI-PVI
Status: Completed | Type: Observational
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Department of Anesthesiology Johannes Gutenberg University Mainz, Department of Anesthesiology Johannes Gutenberg University Mainz
Other Study IDs: AS_001
Record Dates: First submitted 2011-07-05; First posted 2011-07-07 (Estimated); Last update posted 2011-09-07 (Estimated); Status verified 2011-07

CONDITIONS: Perfusion Index and Pleth Variability Index; Interscalene Blocks; Orthopedic Surgery
Keywords: PI; PVI; Interscalene block

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to:

1. To describe effects of interscalene nerve blocks on perfusion index (PI) and pleth variability index (PVI) (Radical 7, Masimo Cooperation, Irvine, CA) before and after induction of general anesthesia.
2. To compare effects of fluid-bolusing on PI and PVI of the anesthetized and non-anesthetized limb.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for shoulder or upper arm surgery
* ASA 1-3
* written informed consent
* approval from the local ethics committee

Exclusion Criteria:

* arrhythmia
* patients suffering from severe vascular disease, coronary artery (CCS IV) disease
* anaemia (haemoglobin < 7mg/dl)
* patients in whom a tidal volume of 8ml/kg cannot be delivered safely

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for surgery of the shoulder and the upper arm.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2010-09

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology, Johannes Gutenberg-University Mainz, Mainz, Rhineland-Palatinate, Germany

REFERENCES:
- [Derived] Sebastiani A, Philippi L, Boehme S, Closhen D, Schmidtmann I, Scherhag A, Markstaller K, Engelhard K, Pestel G. Perfusion index and plethysmographic variability index in patients with interscalene nerve catheters. Can J Anaesth. 2012 Dec;59(12):1095-101. doi: 10.1007/s12630-012-9796-3. Epub 2012 Oct 2. PMID 23055034